CLINICAL TRIAL: NCT07370168
Title: Contact Lens Aftercare Refinement Initiative for Frequency Intervals
Brief Title: Do Daily Disposable Soft Contact Lenses Require Frequent Checks After the Initial Fitting is Complete in Adults Under 40 With No Contraindications
Acronym: CLARIFI
Status: Enrolling by invitation | Type: Observational
Sponsor: Aston University (Other)
Collaborators: CooperVision, Inc. (Industry)
Responsible Party: Principal Investigator, Debarun Dutta, Doctor Senior Lecturer, School of Optometry, Aston University
Other Study IDs: HLS21269
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Healthy Participants
Keywords: Contact Lens; Daily Disposable; Soft; Aftercare

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1- In-person: Receives In-person Scheduled Contact Lens Aftercare
- Cohort 2 - Remote: Receives Telecommunication Scheduled Contact Lens Aftercare

SUMMARY:
Patients who want to wear contact lenses often need to visit the optician multiple times. For example, they might go for an eye test, then return for the contact lens fitting, come back to pick up the lenses, and then again for follow-up care and check-ups. Right now, there are no clear guidelines on how many visits are needed for efficient and high-quality contact lens care.

The purpose of the current study is to understand the scheduling and frequency of follow-up visits required for both new contact lens wearers and those who are experienced.

DETAILED DESCRIPTION:
Overview / Background / unmet need:

Soft contact lens technology and contact lens related clinical practice have evolved significantly over the last three decades[1] . Improvements have been made in every direction: significant improvement in material biocompatibility and transmissibility, enhanced lens designs and optics, wider power ranges, better care regimes, and almost all possible and flexible modalities of lens wear and replacement frequencies. Similarly, eye care professionals (ECPs) are also directed by UK clinical practice guidelines detailed by professional bodies which are aimed at maintaining high levels of ocular health and providing satisfactory vision and comfort [2].

However, current approach for soft contact lens fitting and subsequent follow up appointments, which is defined in the UK by the number of patient visits required to satisfy a new contact lens fit[3], proceeded by follow-up visits to continue safe and healthy lens wear have remained largely conservative[3] . The general course of action has not evolved over recent decades where patients are recalled several times during their journey of contact lens fit in the first few months of wear, likely due to potential complications and challenges faced by the earlier lens materials, designs and limited replacement frequencies [4] and habits formed by ECPs over the years. Although current contact lens materials are superior for benefits such as oxygen performance, wettability and deposition, a variety of wearing modalities and replacement frequencies are available, along with a wide range of powers such that virtually all potential wearers can be fitted with contact lenses. With the advent of a range of virtual assessment tools, contact lens aftercare and frequency of routine clinic visits remained empirical and outdated whether for new or refitting existing contact lens wearers[3] .

Currently, a new soft contact lens wearer may need to visit an ECP several times to finalise a fitting whether for a new or existing wearer, and whether this is a spherical, or toric lens, which can consume significant ECP chair time and may cause patient inconvenience. Given the clinical performance and success rates with contemporary soft contact lenses, and possibility of fitting support with online tools and a range of virtual consultation options, the number of in person visits could be reduced.

The global market in terms of lens replacement in 2023, about half of all lenses prescribed were daily disposables (DD) and one third were monthly replaced contact lenses. In the United Kingdom, more than 60% of contact lens fits were DD which has been steadily increasing over the last few decades [5]. The increase in popularity of DD lenses is also supported by minimised risk of significant and non-significant adverse events related to these lenses, however the absolute rates and risks of microbial keratitis (MK) has remained consistent at 2-4 per 10,000 contact lens wearers per year [6].

Given DD lenses bypass direct dependence on multipurpose care solutions and cases, the matter of patient convenience has also made DD lenses more popular than ever. Patients also have spare lenses available in the event of loss or damage. DD lenses have less chance of spoilation from lens deposits and minimum chance of exposure to pathogenic microorganisms which may lead to microbial adverse events [7]. In addition, a wide range of spherical and toric DD lenses are currently available, which typically range between +8.00 Ds to -12.00Ds, whereas up to 2.25 Dc astigmatic corrections are available. DD contact lens wear is reported to maintain high patient comfort and visual acuity, coupled with the wide range of available parameters underpin high patient comfort and visual satisfaction [8, 9].

Objectives:

Project objective is to evaluate the current provision and frequency of patient follow up visits required for a new or experienced contact lens fit.

A clinical study is proposed to determine the number of follow up appointments required for optimal clinical and satisfactory outcomes in the weeks following a soft contact lens fitting, for both neophytes and existing wearer refits, and investigate delivery of care across different channels such as remote when appropriate.

Endpoints:

* Both patient and ECPs are satisfied and no difference in patient comfort with the number of follow up visits after one year
* A follow up telephone call 2-weeks ± 10 days after initial visit is adequate to maintain safe and effective lens wear for first 1 year of contact lens wear

Study design:

A controlled, open label, 4-arm study will be designed where daily disposable new lens wearers (neophytes) will be assigned into four groups. The study will receive human ethics committee approval and will be registered with a clinical trial registry.

The study will have the following visits (Table 1 for phase-I and table 2 for phase-II) and follow ups scheduled over a duration of 1 year (365 ± 60 days) and will be conducted in support with independent UK practices and those from the Specsavers Group. Coopervision daily disposable spherical and toric lenses will be used. An experienced lens wearer is designated to a participant who has worn lenses more than 3 months in lifetime, anyone with less experience of lens wear is designated as an inexperienced lens wearer (neophytes). Patient satisfaction and comfort will be scored in 1-10 (1 being highly unsatisfied or uncomfortable). Similarly, ECP satisfaction will be graded 1-10 (1 being highly unsatisfied).

Sample size: A total of 65 new contact lens wearers (neophytes) for cohort 1 and 2, and 60 experienced wearers for cohort 3 and 4 will be recruited (Table 1 and 2 respectively), totalling to 250 patients. Calculation was based on identifying significant difference in patient comfort after 1 year of lens wear with 80% power, significance 0.05(G*Power). The dropout rate for experienced contact lens wearers can be up to 25% over 1 year of wear, requiring 60 participants for each cohort. Whereas dropout rates for new contact lens wearers during 1st year can be up to 35% [7], requiring 65 participants.

Table 1 (Phase I) Visit number Control cohort-1 with empirical visits for neophytes (n=65) Test cohort-2 with modified visits for neophytes (n=65) 1.0 Initial assessment and fitting with or without teach and collection of CLs (Day 0) Initial assessment and fitting with or without teach and collection of CLs (Day 0) 1.1 Teaching visit (Day 0+10 days) (unscheduled visit - if required) Teaching visit (unscheduled visit - if required) 2.0 Follow up in office assessment (Day 14 ± 10 days) Follow-up telephone call* (Day 14±10 days) 3.0 Follow up in office assessment (Day 365 ± 60 days)# Follow up in office assessment (Day 365 ± 60 days)# Any additional call/visit will be termed as 'unscheduled visit'. Any visit not within window period will be termed as 'late visit', but all will be recorded.

Table 2. (Phase II) Visit number Control cohort-3 with empirical visits experienced wearers (n=60) Test cohort-4 with modified visits experienced wearers (n=60) 1.0 Initial assessment and fitting with or without teach (Day 0)

Initial assessment and fitting with or without teach (Day 0)

1.1 Teaching and collection if needed (Day 7±4days) Teaching and collection if needed (Day 7±4days) 2.0 Follow up in office assessment (Day 14 ± 10 days following collection of CLs) Follow-up telephone call* (Day 14 ± 10 days following collection of CLs) 3.0 Follow up in office assessment (Day 365 ± 30 days) Follow up in office assessment (Day 365 ± 30 days) Any additional call/visit will be termed as 'unscheduled visit'. Any visit not withing window period will be termed as 'late visit'.

Data collection for each visit will include:

Visit 1.0 and 3.0 (all cohorts):

This will include comprehensive ocular assessments such as: visual acuity, detailed slit lamp assessments for anterior eye, lens fit assessment and ocular comfort (1-10). These are listed below:

* Reason of wear
* General history
* Allergies
* Ocular history
* Contact lens wear history (cohort 3 and 4)
* Occupation / hobbies
* Lens details/parameters
* Best Corrected Visual Acuity (BCVA)
* Detailed slit lamp assessments of anterior eye including Lids /lashes Conjunctiva Limbus Neovascularisation / Oedema Cornea / Staining
* Soft contact lens fitting Parameters HVID Pupil diameter Keratometry/topography Centration and coverage Blink movement Lag Push up test Overall impression/other comments Comfortable with self application and removal - Yes/ No (visit 1.0 only: if teaching included) Other notes
* Patient Comfort (visit 3.0 only, scores 1-10; where 1 highly uncomfortable and 10 very comfortable)
* Patient satisfaction (visit 3.0 only, scores 1-10; where 1 highly uncomfortable and 10 very comfortable)
* Ease of lens handling/application and removal (1-10; 10 being very easy; if teaching is done in visit 1.0)
* Practitioner satisfaction with patient follow ups (visit 3.0 only, scores 1-10; where 1 highly unsatisfied and 10 highly satisfied) Visit 1.1 (all cohorts)
* Teaching of lens application and removal, which will include explaining to the patient about the type, storage, safety and compliance.
* Ease of lens handling/application and removal (1-10; 10 being very easy; if teaching is not done visit 1.0)
* Performed by ECP/someone else Visit 2.0 (cohort 1 and 3 with in person follow ups)
* Reason for visit
* Age of lens / modality / solution (NA for this study/SS might have in clinic form)
* History and symptoms to mirror those for the remote cohort.
* Wear times Hrs/day Days/week
* Vision with lens
* Over refraction
* Final VA
* Lens fitting assessments Centration and coverage Blink movement Lag Push up test Overall impression/other comments
* Detailed slit lamp assessments of anterior eye including Lids /lashes Conjunctiva Limbus Neovascularisation / Oedema Cornea / Staining
* Hours of lens wear/day
* Comfort at the start and end of lens wear: rate 1-10 (10 being highly comfortable)
* Ease of lens handling/application and removal (1-10; 10 being very easy)
* Comfort score 1-10 (1 being very uncomfortable)

  *Visit 2.0 (cohort 2 and 4 clinician led telephone call)
* Greetings and overall wellbeing, check lens specs, any changes in symptoms / experience since last visit (any significant change reported by patient would trigger in person visit)
* Vision with contact lens - rate 1-10 (10 being highly satisfactory) any changes in vision throughout day of wear
* Duration of lens wear (hr) per day / days per week
* Hours of comfortable lens wear per day
* Comfort at the start and end of lens wear: rate 1-10 (10 being highly comfortable)
* Ease of lens handling/application and removal (1-10; 10 being very easy)
* Any significant eye redness, discomfort, discharge, other adverse events, any other issues (yes will trigger in person visits)
* Confirm next follow up and provide contact details for any questions
* Thank you

Inclusion/exclusion criteria:

Inclusion criteria

* Age between 18 to 40 years
* Willing to use the prescribed soft daily disposable contact lenses
* Normal ocular health
* Rx range from +8.00 to -12.00DS and up to 2.50DC (within range that could be fitted by CV 1 day CLs)
* Willing to provide written consent in English
* Can attain good vision: Best-corrected visual acuity of 6/12 or better in each eye
* Have no history of ocular surgery, injury, recent or current infection within the last 3 months
* Have no known allergies to the study products
* Willing to attend the scheduled study visits and adhere to instructions
* If taking fish oil or tear supplements, should have started at least 3 months prior to starting the study and not planned changes to supplement intake during the study Exclusion criteria
* RGP contact lens wear
* Extended contact lens wear
* Re-usable contact lens wear
* Contact lenses for presbyopia correction
* Soft contact lens wear for therapeutic/bandage purposes
* Soft contact lenses for myopia control
* Experienced contact lens wearer with a history of regular lens wear more than 3 months
* Unstable refractive error
* Binocular vision anomaly not controlled by contact lenses
* Patients require Presbyopic correction or age more than 40 years
* Not on a stable medication
* Participation in another clinical trial within 2 weeks of participation in this study
* History or presence of any ocular disorder or condition in either eye that would likely interfere with the interpretation of the study results or patient safety
* Self-reported pregnancy or lactation
* Any ocular or systemic condition that may contradict contact lens wear

Inclusion/exclusion exceptions:

* The investigator has the right to exclude any patient's participation in the study if he/she deems it to be in the best interest of the patient
* Minor exceptions to the inclusion / exclusion criteria will be submitted to, and considered by the PI and approved as required.

Informed consent:

Prior to the screening visit, participants will be provided with an informed consent form and be given the chance to review and ask questions before written informed consent is obtained. The participant will sign and date the informed consent form.

Statistical analysis: Paired-t-test, Repeated measures ANOVA or linear mixed model analysis using Bonferroni adjustment for multiple comparisons and P-value set at p<0.05.

Dissemination plan: sample

1. Presentation at an International conference such as the British Contact Lens Association, UK or American Academy of Optometry, USA.
2. Publication in peer-review journals: Contact Lens and Anterior Eye or Ophthalmic Physiological Optics

Budget:

Funded 50:50 by Coopervision and Aston University

References:

1. Dutta D, Woods CA. Reflection of contact lens practice. Contact lens & anterior eye : the journal of the British Contact Lens Association 2019;42(6):587-9. https://doi.org/10.1016/j.clae.2019.10.003.
2. Sulley A, Young G, Hunt C. Factors in the success of new contact lens wearers. Contact lens & anterior eye : the journal of the British Contact Lens Association 2017;40(1):15-24. https://doi.org/10.1016/j.clae.2016.10.002.
3. Efron N, Morgan PB. Rethinking contact lens aftercare. Clinical & experimental optometry : journal of the Australian Optometrical Association 2017;100(5):411-31.
4. Morgan PB, Efron N. Influence of practice setting on contact lens prescribing in the United Kingdom. Contact lens & anterior eye : the journal of the British Contact Lens Association 2015;38(1):70-2.
5. Morgan et al. International contact lens prescribing trend in 2023. Cont Spectrum. 2024; January(39)20-28.
6. Szczotka-Flynn LB, Shovlin JP, Schnider CM, Caffery BE, Alfonso EC, Carnt NA, Chalmers RL, Collier S, Jacobs DS, Joslin CE, Kroken AR, Lakkis C, Pearlman E, Schein OD, Stapleton F, Tu E, Willcox MDP. American Academy of Optometry Microbial Keratitis Think Tank. Optom Vis Sci. 2021 Mar 1;98(3):182-198.
7. Sulley A, Dumbleton K. Silicone hydrogel daily disposable benefits: The evidence. Cont Lens Anterior Eye. 2020 Jun;43(3):298-307.
8. Maldonado-Codina C, Navascues Cornago M, Read ML, Plowright AJ, Vega J, Orsborn GN, Morgan PB. The association of comfort and vision in soft toric contact lens wear. Cont Lens Anterior Eye. 2021 Aug;44(4):101387.
9. Ichijima H, Karino S, Sakata H, Cavanagh HD. Improvement of Subjective Symptoms and Eye Complications When Changing From 2-Week Frequent Replacement to Daily Disposable Contact Lenses in a Subscriber Membership System. Eye Contact Lens. 2016 May;42(3):190-5.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 to 40 years

* Willing to use the prescribed soft daily disposable contact lenses
* Normal ocular health
* Rx range from +8.00 to -12.00DS and up to 2.50DC (within range that could be fitted by CV 1 day CLs)
* Willing to provide written consent in English
* Can attain good vision: Best-corrected visual acuity of 6/12 or better in each eye
* Have no history of ocular surgery, injury, recent or current infection within the last 3 months
* Have no known allergies to the study products
* Willing to attend the scheduled study visits and adhere to instructions
* If taking fish oil or tear supplements, should have started at least 3 months prior to starting the study and not planned changes to supplement intake during the study

Exclusion Criteria:

* RGP, Extended Wear (re-usable), presbyopic, therapeutic/cosmetic, or myopia control contact lens wear

  * Experienced contact lens wearer with a history of regular lens wear more than 3 months
  * Unstable refractive error
  * Binocular vision anomaly not controlled by contact lenses
  * Patients require Presbyopic correction or age more than 40 years
  * Age < 18 years old
  * Not on a stable medication
  * Participation in another clinical trial within 2 weeks of participation in this study
  * History or presence of any ocular disorder or condition in either eye that would likely interfere with the interpretation of the study results or patient safety
  * Self-reported pregnancy or lactation
  * Any ocular or systemic condition that may contradict contact lens wear ** *The investigator has the right to exclude any patient's participation in the study if he/she deems it to be in the best interest of the patient. Minor exceptions to the inclusion / exclusion criteria will be submitted to, and considered by, the Pl and approved as required. This includes 'drop-outs' that subsequently return to contact lens wear during the study trial.

    * OO/CLO (ECP) Clinical Judgement

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: United Kingdom Specsavers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safe and effective lens wear for first 1 year of contact lens wear | Following Patient for One Year
  Phone Aftercare Adequately Safe and effective

SECONDARY OUTCOMES:
Satisfaction patient comfort with the number of follow up visits after one year | One Year
  Both patient and ECPs are satisfied and no difference in patient comfort with the number of follow up visits after one year

CONTACTS AND LOCATIONS:
Locations (1):
- Specsavers, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Consent has not been given by participants for individual data to be shared